CLINICAL TRIAL: NCT04322968
Title: Low Dose Ketamine Infusion for Comorbid Posttraumatic Stress Disorder and Chronic Pain Patients
Brief Title: Ketamine Infusion for Comorbid PTSD and Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Ann Arbor Healthcare System (U.S. Federal Agency)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-2017-1015
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-11

CONDITIONS: PTSD; Chronic Pain
Keywords: PTSD; chronic pain; ketamine infusion
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Patient with and without PTSD were randomized to receive either ketamine or ketorolac. Single IV infusion of ketamine hydrochloride (0.5 mg/kg) was administered over 40 minutes. Ketorolac 15 mg was reconstituted in 500 cc of normal saline administered over 40 minutes.
Who Masked: Participant, Outcomes Assessor
Masking Description: All study personnel, including rater, patients, and data analysts, were blinded to randomization order. Only the anesthesiologist performing the infusion was not blinded in order to prepare for possible side effects of each medication.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Chronic pain with PTSD+IV ketamine infusion (Experimental)
  Interventions: Drug: A single low dose ketamine infusion as compared to the IV infusion of active placebo - ketorolac on chronic pain and PTSD symptoms.
- Chronic pain with PTSD+IV ketorolac infusion (Active Comparator)
  Interventions: Drug: A single low dose ketamine infusion as compared to the IV infusion of active placebo - ketorolac on chronic pain and PTSD symptoms.
- Chronic pain without PTSD+IV ketamine infusion (Experimental)
  Interventions: Drug: A single low dose ketamine infusion as compared to the IV infusion of active placebo - ketorolac on chronic pain and PTSD symptoms.
- Chronic pain without PTSD+IV ketorolac infusion (Active Comparator)
  Interventions: Drug: A single low dose ketamine infusion as compared to the IV infusion of active placebo - ketorolac on chronic pain and PTSD symptoms.

INTERVENTIONS:
Drug: A single low dose ketamine infusion as compared to the IV infusion of active placebo - ketorolac on chronic pain and PTSD symptoms. — Subjects were randomized into 4 treatment groups: chronic pain subjects treated with ketorolac, chronic pain subjects treated with ketamine, chronic pain+PTSD subjects treated with ketorolac, and chronic pain+PTSD subjects treated with ketamine.

SUMMARY:
The purpose of the study is to investigate the effectiveness of low dose IV ketamine infusion in the treatment of patients with PTSD and comorbid chronic pain.

Hypothesis: A single ketamine infusion should be associated with significantly greater reduction in core PTSD symptom levels after the treatment and such an effect is not only due to its analgesic properties but also through unknown mechanism of action that maybe related to NMDA/AMPA receptor modulation.

DETAILED DESCRIPTION:
To date, treatment options (i.e. psychotherapy, antidepressant medications) for patients with PTSD, are relatively few, and considering their limited efficacy, novel therapies have gained interest among researchers and treatment providers alike. Among patients with chronic pain about one third suffer from comorbid PTSD, which further complicates their already challenging pharmacological regimens. Low dose ketamine infusion has shown promise in PTSD, and in treatment of chronic pain, however they have not been studied in comorbid population and under rigorous control conditions. The investigators compared the effects of a single dose of either ketamine (0.5 mg/kg) or ketorolac (15 mg) over a 40-minute of IV infusion in chronic pain patients with and without PTSD, in double blind, randomized study. Measures were collected before, during, 1 day and 7 days after the infusion.

ELIGIBILITY:
Inclusion Criteria:

Veterans with chronic pain as defined by having any chronic pain beyond 6 months in duration with and without PTSD diagnoses (participants must meet DSM-V criteria for current post-traumatic stress disorder (PTSD) and have received a diagnosis of PTSD greater than or equal to 3 months prior to assessment); they also will be either free of concomitant use of psychotropic and/or pain medications for at least 6 weeks or on stable doses of those medications within the last 6 weeks prior to randomization and for the duration of the study; if applicable, current frequency and duration of psychotherapy sessions must remain stable for at least 6 weeks prior to beginning of the study.

Exclusion Criteria:

Inability to speak English, inability or unwillingness to provide written informed consent; moderate-to-severe cognitive impairment (Mini-Mental State Examination scores<20 administered by a trained clinician); current or lifetime history of psychotic or bipolar disorder; current bulimia or anorexia nervosa, alcohol abuse or dependence in the previous 3 months; serious unstable medical illness or sleep apnea; HTN, prolonged QT interval, peptic ulcer disease or recent history of GI-bleed, renal insufficiency, active substance use disorder, active suicidal or homicidal ideation on presentation; pregnancy (confirmed by baseline lab test), the initiation of female hormonal treatments within 3 months of screening, or inability or unwillingness to use a medically accepted contraceptive method for the duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ann Arbor VA Medical Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Local IRB has conducted informed consent audit for the study and the investigators have been compliant with it.

REFERENCES:
- [Background] Asmundson GJ, Bonin MF, Frombach IK, Norton GR. Evidence of a disposition toward fearfulness and vulnerability to posttraumatic stress in dysfunctional pain patients. Behav Res Ther. 2000 Aug;38(8):801-12. doi: 10.1016/s0005-7967(99)00101-1. PMID 10937428
- [Background] Kessler RC, Chiu WT, Demler O, Merikangas KR, Walters EE. Prevalence, severity, and comorbidity of 12-month DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):617-27. doi: 10.1001/archpsyc.62.6.617. PMID 15939839
- [Background] Feder A, Parides MK, Murrough JW, Perez AM, Morgan JE, Saxena S, Kirkwood K, Aan Het Rot M, Lapidus KA, Wan LB, Iosifescu D, Charney DS. Efficacy of intravenous ketamine for treatment of chronic posttraumatic stress disorder: a randomized clinical trial. JAMA Psychiatry. 2014 Jun;71(6):681-8. doi: 10.1001/jamapsychiatry.2014.62. PMID 24740528
- [Background] Albott CS, Lim KO, Forbes MK, Erbes C, Tye SJ, Grabowski JG, Thuras P, Batres-Y-Carr TM, Wels J, Shiroma PR. Efficacy, Safety, and Durability of Repeated Ketamine Infusions for Comorbid Posttraumatic Stress Disorder and Treatment-Resistant Depression. J Clin Psychiatry. 2018 May/Jun;79(3):17m11634. doi: 10.4088/JCP.17m11634. PMID 29727073
- [Background] Sigtermans MJ, van Hilten JJ, Bauer MCR, Arbous SM, Marinus J, Sarton EY, Dahan A. Ketamine produces effective and long-term pain relief in patients with Complex Regional Pain Syndrome Type 1. Pain. 2009 Oct;145(3):304-311. doi: 10.1016/j.pain.2009.06.023. Epub 2009 Jul 14. PMID 19604642
- [Background] Noppers I, Niesters M, Swartjes M, Bauer M, Aarts L, Geleijnse N, Mooren R, Dahan A, Sarton E. Absence of long-term analgesic effect from a short-term S-ketamine infusion on fibromyalgia pain: a randomized, prospective, double blind, active placebo-controlled trial. Eur J Pain. 2011 Oct;15(9):942-9. doi: 10.1016/j.ejpain.2011.03.008. Epub 2011 Apr 11. PMID 21482474

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Pain With PTSD+IV Ketamine Infusion; Chronic Pain Without PTSD+IV Ketamine Infusion: A single low dose iv ketamine infusion (0.5 mg/kg) administered over 40 min.
- Chronic Pain With PTSD+IV Ketorolac Infusion; Chronic Pain Without PTSD+IV Ketorolac Infusion: A single iv infusion of ketorolac (15 mg) administered over 40 min.
Period: Overall Study
Arm/Group | Chronic Pain With PTSD+IV Ketamine Infusion | Chronic Pain With PTSD+IV Ketorolac Infusion | Chronic Pain Without PTSD+IV Ketamine Infusion | Chronic Pain Without PTSD+IV Ketorolac Infusion
Started | 11 | 10 | 10 | 10
Completed | 10 | 9 | 10 | 10
Not Completed | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Pain With PTSD+IV Ketamine Infusion | Chronic Pain With PTSD+IV Ketorolac Infusion | Chronic Pain Without PTSD+IV Ketamine Infusion | Chronic Pain Without PTSD+IV Ketorolac Infusion | Total
Number analyzed (Participants) | 10 | 9 | 10 | 10 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 10 | 10 | 39
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 1 | 1 | 9
  Male | 6 | 6 | 9 | 9 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 8 | 9 | 10 | 37
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 9 | 10 | 10 | 39

OUTCOME MEASURES:

1. Primary Outcome: Impact of Event Scale-Revised (IES-R)
Description: Severity of PTSD symptoms; items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The IES-R yields a total score (ranging from 0 to 88); higher scores mean worse symptoms
Time Frame: 24 hrs post-infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Pain With PTSD+IV Ketamine Infusion | Chronic Pain With PTSD+IV Ketorolac Infusion | Chronic Pain Without PTSD+IV Ketamine Infusion | Chronic Pain Without PTSD+IV Ketorolac Infusion
Number analyzed (Participants) | 10 | 9 | 10 | 10
units on a scale | 36.33333333 (17.27715254) | 37 (15.77973384) | 10.44444444 (14.34495653) | 15.64705882 (17.05484233)

2. Primary Outcome: Visual Analogue Scale (VAS)
Description: Severity of chronic pain symptoms; using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100; a higher score indicates greater pain intensity.
Time Frame: 24 hrs post-infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Pain With PTSD+IV Ketamine Infusion | Chronic Pain With PTSD+IV Ketorolac Infusion | Chronic Pain Without PTSD+IV Ketamine Infusion | Chronic Pain Without PTSD+IV Ketorolac Infusion
Number analyzed (Participants) | 10 | 9 | 10 | 10
units on a scale | 37.22222222 (24.69705336) | 49.66666667 (23.44141634) | 29.88888889 (24.15286962) | 38.70588235 (28.12197696)

3. Secondary Outcome: Impact of Event Scale-Revised (IES-R)
Description: as for outcome 1
Time Frame: 1 week post-infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Pain With PTSD+IV Ketamine Infusion | Chronic Pain With PTSD+IV Ketorolac Infusion | Chronic Pain Without PTSD+IV Ketamine Infusion | Chronic Pain Without PTSD+IV Ketorolac Infusion
Number analyzed (Participants) | 10 | 9 | 10 | 10
units on a scale | 28.22 (22.60) | 33.66666667 (20.43281674) | 11.44 (17.47) | 13.41 (16.84)

4. Secondary Outcome: Visual Analogue Scale (VAS)
Description: as for outcome 2
Time Frame: 1 week post-infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Pain With PTSD+IV Ketamine Infusion | Chronic Pain With PTSD+IV Ketorolac Infusion | Chronic Pain Without PTSD+IV Ketamine Infusion | Chronic Pain Without PTSD+IV Ketorolac Infusion
Number analyzed (Participants) | 10 | 9 | 10 | 10
units on a scale | 48.22 (31.59) | 52.88 (21.55) | 43.33 (19.28) | 48.23 (21.72)

5. Secondary Outcome: Brief Pain Inventory (Short Form)
Description: Severity of pain, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours or the past week; No scoring algorithm, but "worst pain" or the arithmetic mean of the four severity items can be used as measures of pain severity (a range of 0-10, with 10 being worse scores); the arithmetic mean of the seven interference items can be used as a measure of pain interference (a range of 0-10, with 10 being worse scores). The total score is reported for severity items and interference items, which range from 0-40 and 0-70, respectively. Higher values represent worse outcome.
Time Frame: 1 week post-infusion
Population: BPI- pain scale and pain interference
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chronic Pain With PTSD+IV Ketamine Infusion | Chronic Pain With PTSD+IV Ketorolac Infusion | Chronic Pain Without PTSD+IV Ketamine Infusion | Chronic Pain Without PTSD+IV Ketorolac Infusion
Number analyzed (Participants) | 10 | 9 | 10 | 10
units on a scale
  Pain interference Scale | 38.62 (24.03) | 25.66 (20.32) | 9.62 (7.44) | 28.33 (21.96)
  Pain severity Scale | 20.75 (10.55) | 14.66 (9.53) | 12.75 (5.44) | 22.66 (9.13)

6. Other Pre Specified Outcome: Patient-Rated Inventory of Side Effects (PRISE20)
Description: Patient self report used to qualify side effects by identifying and evaluating the tolerability of each symptoms; 20 items; higher scores mean worse side effects
Time Frame: baseline-1 week post-infusion
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Clinician-Administered Dissociative States Scale (CADSS)
Description: Dissociative, psychotomimetic, and manic symptoms; 27-item scale with 19 subject-rated items and 8 items scored by an observer; higher scores mean worse present-state dissociative symptomatology
Time Frame: baseline-1 week post-infusion
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Chronic Pain With PTSD+IV Ketamine Infusion | Chronic Pain With PTSD+IV Ketorolac Infusion | Chronic Pain Without PTSD+IV Ketamine Infusion | Chronic Pain Without PTSD+IV Ketorolac Infusion
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT04322968/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT04322968/SAP_001.pdf